CLINICAL TRIAL: NCT07291674
Title: Predictors and Outcome of Rupture Hepatocellular Carcinoma in Assuit Unversity Hospitals
Brief Title: Predictors and Outcome of Rupture HCC in AU Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mokhtar Omar Khaled, Principle investigator, Assiut University
Other Study IDs: Rupture HCC in AU hospitals
Record Dates: First submitted 2025-09-28; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HCC Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aime of the study is To identify the Prevalence of rupture of HCC among patients diagnosed with HCC at Assiut University Hospitals in the last five years.

,detect the Risk factors and predictors of rupture HCC. and identify the survival rate in 1 year post rupture HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* *Age ≥18 years

  * Diagnosed with HCC (radiologically or histopathologically)
  * Evidence of spontaneous rupture confirmed by imaging or surgical exploration
  * Admitted to the hospital during the study period

Exclusion Criteria:

* * Traumatic liver rupture

  * Non-HCC liver malignancies
  * Incomplete medical records or missing imaging data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years) with a confirmed diagnosis of HCC and evidence of spontaneous tumor rupture will be included. Rupture will be defined radiologically (via CT scan or ultrasound showing hemoperitoneum and liver lesion discontinuity) or confirmed intraoperatively
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Detect Prevalence of rupture of HCC among patients diagnosed with HCC at Assiut University hospitals in the last five years. | Baseline
  The following variables will be extracted:
  1. Demographic data (age, gender, residence)
  2. Liver disease history (HBV/HCV status, Child-Pugh score, MELD score)
  3. Tumor characteristics (size, number, location, vascular invasion)
  4. Clinical presentation (abdominal pain, hypotension, hemoglobin level)
  5. Diagnostic imaging findings (CT, ultrasound)
  6. Management approach (conservative, transarterial embolization [TAE], surgical resection)

CONTACTS AND LOCATIONS:
Overall Officials: Mokhtar Qaleed, Principal Investigator — Assiut University; Mahmoud Ashri, Study Director — Assiut University; Bahaa Osman Taha, Study Director — Assiut University